# Cover page with the Official Title of the study:

An Internet-based ,Self-applied Treatment of Rat Phobia using a Virtual Therapist Assistant: Study Protocol for a Randomized Controlled Trial. Date: October 4, 2021









### Informed consent

A group of researchers from the Universidad Autónoma de Baja California (UABC), Universidad Nacional Autónoma de México (UNAM), Tecnológico Nacional de México campus Instituto Tecnológico de Ensenada (TecNM/ITE), and the Universidad Internacional de Valencia (VIU), are conducting a study in order to implement and validate an online intervention based on exposure therapy through a virtual therapeutic assistant called Thera, that interacts verbally with the patient to guide and control exposure therapy for phobias to animals delivered through several channels. Thera also analyzes the physiological records (heart rate) of the patient in real-time to determine their emotional state during the intervention.

The content of the intervention will be self-applied through a web application including the guidance of Thera. In order to integrate the benefits that Internet-based interventions could provide and the assistance of a virtual therapist to guide and personalize the progress of the treatment according to the user. The results of this research will be analyzed for research purposes and, therefore, they can be published in journals, scientific books or disseminated by other means to the scientific community, taking care at all times of the confidentiality and anonymity of the data of the participants. This study has the approval of the Research Ethics Committee, from the Universidad Autónoma de Baja California. Approval date June 8<sup>th</sup>, 2021. Identification number: POSG/021-1-03. It is important to mention that you will not be asked for any sensitive data or your name, in addition to the fact that the intervention will always be completely free.

#### Exclusion criteria:

- 1. Receive another type of psychological or psychopharmacological treatment.
- 2. Being diagnosed with another type of anxiety disorder or some psychopathology.
- 3. Present any medical condition that puts your life at risk (heart disease, respiratory disease, pregnancy, among others).

#### The instruments to answer are:

- 1. Fear scale.
- 2. Anxiety scale.
- 3. Sense of presence and judgment of reality.
- 4. User's satisfaction.
- 5. Perception of utility and ease of use.
- 6. Patient improvement scale.

If you agree with what is proposed, please click on accept, otherwise you can close your internet window. In this application, you indicate that you agree to voluntarily participate in this research that we are conducting and, therefore, willing/complete the questionnaires.

## Procedure:

- If you are willing to participate in the study, we will ask you to sign that you are interested in participating.
- The confidentiality of the information you provide us will be taken care of at all times. These activities will be carried out by an associate student and supervised by the researchers indicated in the confidentiality commitment found at the end of this document.
- You can do the activity at a time and day that does not interfere with your main activities.
- You are free to withdraw from the assessment at any time.

• The activities carried out during this study do not contain religious, political or ideological information.

# **Benefits:**

If you agree to participate, you will benefit from a free intervention that aims to reduce your symptoms manifested by phobia, thus improving your quality of life. Additionally, you will be notified when, according to the observations, a more extensive assessment process or some other specialized medical or neuropsychological care service is required.

For more questions, you can contact us by mail at <a href="mmeza@uabc.edu.mx">mmeza@uabc.edu.mx</a> or the main researcher of this study, Dr. María Victoria Meza Kubo.

I declare to tell the truth, that i do not have any of the exclusion criteria mentioned above, releasing researchers from any eventuality that may occur during the intervention and I freely agree to participate in the study:

Date: